CLINICAL TRIAL: NCT06039150
Title: Medical Doctor of Anesthesiology and Reanimation
Brief Title: Modified Thoracoabdominal Nerve Block(M-TAPA) in Pediatric Laparoscopic Appendectomies
Acronym: M-TAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ELA ERTEN, Medical Doctor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GULHANEELAERTEN
Record Dates: First submitted 2023-09-03; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain; Laparoscopic Surgery; Pediatrics; Regional Anesthesia; Local Anesthetic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-TAPA group (Experimental): The group to be administered 0.025% Bupivacaine by the anesthesiologist bilaterally in M-TAPA block with a maximum dose of 2 mg/kg before extubation.
  Interventions: Procedure: M-TAPA Block
- LAİ group (Active Comparator): The group to be divided and administered 0.025% Bupivacaine with a maximum dose of 2 mg/kg by the surgeon to 3 port entry sites before extubation
  Interventions: Procedure: Local anesthetic infltration to port sites

INTERVENTIONS:
Procedure: M-TAPA Block — M-TAPA Block; The block will be done by the same experienced anesthesiologist by using ultrasound(USG) after the surgical intervention is completed.The external oblique, internal oblique, and transversus abdominis muscles were shown on the costochondral angle in the sagittal plane at the 10th costal margin by using a high-frequency linear probe. Bilaterally in the midclavicular line at the level of the 10th rib (arcus costarum),0,5 ml/kg 0.25% Bupivacaine (maximum dose 2mg/kg) was administered to between the upper fascia of the transversus abdominis muscle and the lower fascia of the costochondral tissue.
  Arms: M-TAPA group
Procedure: Local anesthetic infltration to port sites — Local anesthetic infiltration to port sites; The surgeon infiltrated 0.5 ml/kg of 0.25% Bupivacaine (maximum dose of 2mg/kg) in the skin, subcutaneous tissue, and muscle fascia at each of the three laparoscopic port areas at the end of the surgery.
  Arms: LAİ group

SUMMARY:
To compare the effect of M-TAPA block and port-site local anesthetic infiltration on postoperative pain in pediatric laparoscopic appendectomies. The main questions it aims to answer are:

* Is M-TAPA block more effective in reducing pain?
* How M-TAPA block affects the use of rescue analgesics in the postoperative period? Participants will have the same anaesthetic agents during surgery, before extubation they will have same analgesic agent for postoperative pain. Participants in the M-TAPA group will undergo USG-guided M-TAPA block bilaterally with % 0.025 Bupivacaine max dose of 2 mg/kg by the same experienced anesthesiologist before extubation. Participants in the LAI group will be administered 0.025% Bupivacaine at a maximum dose of 2mg/kg divided equally and administered by the surgeon at 3 port entry sites before the patient is extubated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American society of Anesthesiologists (ASA) physical status I-II,
* Patients which will undergo Laparoscopic appendectomy due to the diagnosis of acute appendicitis,
* Patients whose parents or legal heirs have consented to participate in the study

Exclusion Criteria:

* Patients with Society of Anesthesiologists (ASA) III-IV status,
* Patients whose parents or legal heirs' disapproval,
* Patients inability to cooperate,
* Patients who have allergy to any of the medications used in the study,
* Patients with perforated appendix
* When the Laparoscopic surgery returns to open shape

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-10-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Total number of rescue analgesic applications | Postoperative first 24 hours
  During the first 24 hours postoperatively, patients' pain will be monitored by Visual Analogue Scale (VAS) scoring. Paracetamol will be given intravenously at a dose of 10mg/kg if the VAS is greater than 4 in pain assessment in the postoperative period. We will record the number of times the patient received rescue analgesics over a 24-hour period.

SECONDARY OUTCOMES:
Comparison of pain between 2 groups in the postoperative period | Postoperative first 24 hours
  The Visual Analogue Scale (VAS) scores were recorded postoperatively at 0 (PACU), 1, 4, 6, 12, and 24 h.
  Visual Analogue Scale (VAS)
  Scale vertical or horizontal from a 10 cm long line drawn as is formed. At the two ends of this line are the two end descriptor word (0 = "no pain at all", 10 = worst/unbearable pain").The patient is asked to place a mark in the appropriate place for the intensity of the pain.

OTHER OUTCOMES:
Comparison of postoperative complications | Postoperative first 24 hours
  Patients will be followed up for 24 hours postoperatively for complications including nausea and vomiting and shoulder pain. And it will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ELA ERTEN, Principal Investigator — Anesthesiology and Reanimation department
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandeman DJ, Bennett M, Dilley AV, Perczuk A, Lim S, Kelly KJ. Ultrasound-guided transversus abdominis plane blocks for laparoscopic appendicectomy in children: a prospective randomized trial. Br J Anaesth. 2011 Jun;106(6):882-6. doi: 10.1093/bja/aer069. Epub 2011 Apr 18. PMID 21504934
- [Background] Ozen V, Acik ME, Ozen N. The modified thoracoabdominal nerve block for post-operative analgesia in paediatric laparoscopic cholecystectomy. J Minim Access Surg. 2024 Oct 1;20(4):452-455. doi: 10.4103/jmas.jmas_174_22. Epub 2023 May 10. PMID 37282431